CLINICAL TRIAL: NCT06183840
Title: OMEGA Trial: A Multicenter Randomized Controlled Non-inferiority Trial of Only MEsh Fixation With a Glue Applicator Comparing Traumatic vs Atraumatic Fixation of the Mesh in Ventral/Incisional Laparoscopic Repair
Brief Title: Only Mesh Fixation With Glue of Ventral/Incisional Laparoscopic Hernia Repair
Acronym: OMEGA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Catala de Salut (Other Government)
Responsible Party: Principal Investigator, Rafael Villalobos Mori, Head of Abdominal Wall Unit Surgery, Institut Catala de Salut
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rafael Villalobos
Record Dates: First submitted 2023-11-06; First posted 2023-12-28 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Ventral Incisional Hernia
Keywords: Ventral hernia; Incisional hernia; Mesh; Glue; Tackers; IPOM plus
MeSH Terms: conditions — Hernia, Ventral; Incisional Hernia

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): Patients with a traumatic fixation of the mesh
  Interventions: Device: Conventional
- Glutack (Experimental): Patient with Glutack mesh fixation
  Interventions: Device: Glutack

INTERVENTIONS:
Device: Glutack — Three ports are used (1x11 mm and 2x5 mm) and after adhesiolysis and the field prepared, the defect is measured with a local standard in a craneo-caudal and transversal directions. Then, the defect is closed with a 2-0 caliber barbed suture following its biggest axis. A Dynamesh IPOM previously hydrated (2-3 min) is introduced throughout the 11mm trocar and extended. After this maneuver, mesh fixation is performed depending on the randomized arm: Glutack
  Arms: Glutack
Device: Conventional — Three ports are used (1x11 mm and 2x5 mm) and after adhesiolysis and the field prepared, the defect is measured with a local standard in a craneo-caudal and transversal directions. Then, the defect is closed with a 2-0 caliber barbed suture following its biggest axis. A Dynamesh IPOM previously hydrated (2-3 min) is introduced throughout the 11mm trocar and extended. After this maneuver, mesh fixation is performed depending on the randomized arm: Traumatic fixation
  Other Names: Traumatic fixation
  Arms: Conventional

SUMMARY:
This multicenter randomized controlled non-inferiority trial of only mesh fixation with a glue applicator is a trial to evaluate the outcomes between atraumatic laparoscopic mesh fixation with GLUTACK-Glubran2® and conventional traumatic fixation, so the primary endpoint of the study is to analyze the recurrence on ventral or incisional hernia repair 2 years postoperatively assessed by a clinical and/or imaging technique.

DETAILED DESCRIPTION:
Patients older than 18 years undergoing an elective ventral/incisional hernia laparoscopic repair with a hernia defect between 4-10cm of transversal defect The patients included are adults with a BMI lesser than 35 Kg/m2 undergoing an elective laparoscopic primary ventral or incisional hernia repair with a fascial transverse defect between 4-8 cm (W2 EHS) on anterior or lateral location (M1-M5 up to 10 cm of length or L1-3) For the interventional procedure, three ports are used (1x11 mm and 2x5 mm) and after adhesiolysis and the field prepared, the defect is measured with a local standard in a craneo-caudal and transversal directions. Then, the defect is closed with a 2-0 caliber barbed suture following its biggest axis. A Dynamesh IPOM previously hydrated (2-3 min) is introduced throughout the 11mm trocar and extended. After this maneuver, mesh fixation is performed depending on the randomized arm (125 per arm): either traumatic fixation with the conventional procedure and device or with Glutack-Glubran®2.

After two years of follow-up, the recurrence will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* All adults with a BMI lesser than 35 Kg/m2 undergoing an elective laparoscopic primary ventral or incisional hernia repair with a fascial transverse defect between 4-8 cm (W2 EHS) on anterior or lateral location (M1-M5 up to 10 cm of length or L1-3)
* ASA grade from I-II
* Informed consent signed

Exclusion Criteria:

* Patients less than 18 years and over 80 years of age.
* Fascial transverse defect less than 4 cm and more than 8 cm.
* Recurrent ventral or incisional hernia in the same place
* Emergency surgery
* Procedure involving concomitant surgeries (e.g. gastrointestinal, biliary or genitourinary surgery)
* BMI greater than 35 Kg/m2
* ASA III-IV
* Pregnancy
* Tobacco

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-03-10 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of the recurrence on ventral or incisional hernia repair 2 years postoperatively assessed by a clinical and/or imaging technique. | 2 years
  The fixation of the mesh with atraumatic material with glue is as good as the conventional traumatic fixation

SECONDARY OUTCOMES:
Rate of postoperative pain between atraumatic and traumatic fixation of the mesh (EuraHS Quality of life scale: 0-10). Ten is the worst outcome | 2 years
Types of comorbidities related on the surgery as visceral adhesions, seroma, hematoma, bulging, port site incisional hernia, recurrence | 2 years
Quality of life (QoL) between the two types of fixations with the EuraHS scale at 1 month, 6 months, 12 months, and 24 months. EurasHS scale of 10 is the worst outcome | 2 years